CLINICAL TRIAL: NCT00467961
Title: Selective Depletion of Alloreacting T Cells Using a Photodepletion Technique to Prevent GVHD After HLA-Matched Peripheral Blood Stem Cell Transplantation for Subjects With Hematologic Malignancies
Brief Title: Stem Cell Transplantation for Patients With Cancers of the Blood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070136; 07-H-0136 (Other: NIH National Heart, Lung and Blood Institute)
Record Dates: First submitted 2007-04-28; First posted 2007-05-01 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2014-12

CONDITIONS: CML (Chronic Myelogenous Leukemia); CLL (Chronic Lymphocytic Leukemia); AML (Acute Myelogenous Leukemia); Acute Lymphocytic Leukemia; MDS (Myelodysplastic Syndrome)
Keywords: CML (Chronic Myelogenous Leukemia); CLL (Chronic Lymphocytic Leukemia); AML (Acute Myelogenous Leukemia); Leukemia; Chronic Lymphocytic Leukemia; CLL; Chronic Myelogenous Leukemia; CML; Acute Myelogenous Leukemia; AML; Acute B-Lymphoblastic Leukemia; ALL; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: Evaluation of selective depletion of alloreactive T cells to prevent graft vs host disease
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Miltenyi system transplant recipients (Experimental): Subjects will receive a myeloablative conditioning regimen of cyclophosphamide, fludarabine and total body irradiation, followed by an infusion of a stem cell product prepared using the Miltenyi CliniMacs system for CD34 selection and a lymphocyte product that has been selectively depleted using the photodepletion approach. Older subjects will receive a lower dose of irradiation to reduce the regimen intensity. Determine appropriate level of post transplant immunosuppression
  Interventions: Combination Product: Miltenyi system

INTERVENTIONS:
Combination Product: Miltenyi system — Subjects will receive a myeloablative conditioning regimen of cyclophosphamide, fludarabine and total body irradiation, followed by an infusion of a stem cell product prepared using the Miltenyi CliniMacs system for CD34 selection and a lymphocyte product that has been selectively depleted using the photodepletion approach.

SUMMARY:
This study will try to improve the safety and effectiveness of stem cell transplant procedures in patients with cancers of the blood. It will use a special machine to separate immune cells (T cells) from the blood of both the donor and the patient and will use photodepletion, a laboratory procedure that selectively kills cancer cells exposed to light. These special procedures may reduce the risk of graft-versus-host-disease (GVHD), a serious complication of stem cell transplants in which the donor's immune cells destroy the patient's healthy tissues, and at the same time may permit a greater graft-versus-leukemia effect, in which the donated cells fight any residual tumor cells that might remain in the body.

Patients between 18 and 75 years of age with a life-threatening disease of the bone marrow (acute or chronic leukemia, myelodysplastic syndrome, or myeloproliferative syndrome) may be eligible for this study. Candidates must have a family member who is a suitable tissue match.

DETAILED DESCRIPTION:
Peripheral blood stem cell transplant research carried out by the NHLBI BMT Unit focus on approaches in transplant techniques designed to decrease graft versus host disease (GVHD), increase the graft-versus-leukemia (GVL) effect, and/or reduce the risk for post-transplant graft rejection or disease relapse.

Ex vivo selective depletion of alloreacting T cells, hereafter referred as selective depletion (SD), represents a translational strategy aiming to reduce severe GVHD whilst preserving GVL. We found that selectively depleted transplants are safe to administer and associated with less severe acute GVHD. This protocol is designed to evaluate the safety and efficacy of photodepletion (PD) as an improved selective depletion procedure in the HLA-matched peripheral blood stem cell transplant setting and to determine whether post-transplant immunosuppression with cyclosporine is necessary to prevent severe GVHD after a photodepleted transplant.

The protocol will accrue subjects ages 18-75 who are diagnosed with a hematological malignancy where allogeneic stem cell transplantation from an HLA-matched sibling would be normally indicated. Diagnostic categories will include acute and chronic leukemias, myelodysplastic syndromes, B-cell lymphomas, multiple myeloma, and myeloproliferative syndromes.

Participants have a central intravenous (IV) line placed into a large vein. The tube is used for giving the donated stem cells and antibiotics and other medicines, for transfusions of red blood cells and platelets, and for collecting blood samples. Treatment starts with a conditioning regimen of chemotherapy (fludarabine and cyclophosphamide) and total body irradiation to suppress immunity and prevent rejection of the donated stem cells. The day after chemotherapy ends, the stem cells are given through the central line. This is followed by transfusion of the donor's immune cells, which have been treated to remove cells that could cause severe GVHD. Also to minimize the risk of GVHD, patients are given cyclosporine. Not all participants receive the same amount of this drug; in order to determine how much immunosuppression is needed to protect against severe GVHD, the length of treatment with cyclosporine varies among patients, depending on when they entered the study and how well preceding patients did.

The average hospital stay for stem cell transplantation is 3 to 4 weeks. Patients return for frequent follow-up visits for the first 2 to 4 months after transplantation. The patient's referring physician is asked to send results of any laboratory testing to the NIH researchers at least every 3 months for the first 3 years and annually thereafter. Patient follow-up visits are scheduled at NIH at 1, 2, and 3 years after transplantation. After 3 years, participants are offered the opportunity to enroll in NHLBI's long-term evaluation and follow-up care protocol.

Subjects will receive a myeloablative conditioning regimen of cyclophosphamide, fludarabine and total body irradiation, followed by an infusion of a stem cell product prepared using the Miltenyi CliniMacs system for CD34 selection and a lymphocyte product that has been selectively depleted using the photodepletion approach (Kiadis Pharma). Older subjects will receive a lower dose of irradiation to reduce the regimen intensity.

To determine appropriate level of post transplant immunosuppression, we will utilize a three sequential de-escalation stage design involving 17 subjects per cohort (minimum 17, maximum 51 total evaluable subjects in study). Stopping rules for non-relapse mortality in each cohort will determine whether to continue to the next stage; to continue accumulating subjects at the same level; or to stop the protocol.

Cohort 1: Low dose cyclosporine until day 90 then dose tapered to stop within 2 weeks.

Cohort 2: If no severe GVHD is encountered in Cohort 1, the cyclosporine withdrawal will begin on day 45.

Cohort 3: If no severe GVHD is encountered in Cohort 2, cyclosporine will not be used in the post-transplant period.

Primary endpoints will be the incidence of acute grade III/IV GVHD at day 90. Secondary endpoints will be standard transplant outcome variables: toxicity, non relapse mortality and survival.

ELIGIBILITY:
INCLUSION CRITERIA:

Recipient Criteria:

* Diagnosed with one of the following hematological conditions:
* Chronic myelogenous leukemia (CML): chronic phase who have failed treatment with imatinib, have intolerance to imatinib, or who did not receive imatinib at therapeutic doses within the first 12 months from diagnosis; accelerated phase or blast transformation.
* Acute B-lymphoblastic leukemia (B-ALL): any of these categories: B-ALL in first remission with high-risk features (presenting leukocyte count greater than 100,000/cu mm, Karyotypes t9; 22, t4, t19, t11, biphenotypic leukemia), all second or subsequent remissions, primary induction failure, partially responding or untreated relapse.
* Acute myelogenous leukemia (AML): AML in first remission - except AML with good risk karyotypes: AML M3 (t15; 17), AML M4Eo (inv 16), AML t (8; 21). All AML in second or subsequent remission, primary induction failure and resistant relapse.
* Myelodysplastic syndromes (MDS): any of these categories - refractory anemia with transfusion dependence, refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia, atypical MDS/myeloproliferative syndromes.
* Myeloproliferative disorders including atypical (Ph negative) chronic myeloid and neutrophilic leukemias, progressing myelofibrosis, and polycythemia vera, essential thrombocythemia in transformation to acute leukemia or with progressive transfusion requirements or pancytopenia.
* Chronic lymphocytic leukemia refractory to fludarabine treatment and with bulky progressive disease or with thrombocytopenia (less than or equal to 100,000 /microl) or anemia (less than or equal to 10g/dl) not due to recent chemotherapy.
* Non-Hodgkin's lymphoma including Mantle cell lymphoma relapsing or refractory to standard of care treatments.
* Multiple myeloma, Waldenstroms macroglobulinemia, unresponsive or relapsed following standard of care treatments.
* Ages 18-75 years inclusive.
* HLA identical (6/6) related donor.
* Ability to comprehend the investigational nature of the study and provide informed consent.

Donor Criteria:

* Related HLA identical (6/6) with recipient.
* Weight greater than or equal to 18 kg.
* Age greater than or equal to 2 or less than or equal to 80 years old.
* For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA:

Recipient Criteria (any of the following):

* Malignant cells expressing a T cell phenotype (in particular T-ALL and T cell NHL).
* DLCO less than 65 percent predicted.
* Left ventricular ejection fraction less than 40 percent (evaluated by ECHO) or less than 30 percent (evaluated by MUGA).
* AST/SGOT greater than 10 times ULN (CTCAE grade IV v3.0).
* Bilirubin greater than 5 times ULN (CTCAE grade IV v3.0).
* Creatinine greater than 4.5 times ULN (CTCAE grade IV v 3.0).
* HIV positive (Recipients who are positive for hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-1/II) are not excluded from participation).
* Positive pregnancy test for women of childbearing age.
* Prior allogeneic stem cell transplantation.
* Estimated probability of surviving less than three months.
* Major anticipated illness or organ failure incompatible with survival from transplant.
* Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and informed consent impossible.

Donor Criteria (any of the following):

* Pregnant or lactating.
* Unfit to receive filgrastim (G-CSF) and undergo apheresis (abnormal blood counts, history of stroke, uncontrolled hypertension).
* Sickling hemoglobinopathies including HbSS, HbAS, HbSC.
* HIV positive Donors who are positive for hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-I/II) will be used at the discretion of the investigator following counseling and approval from the recipient.
* Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the donation of stem cells unlikely and informed consent impossible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minocher M Battiwalla, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Appelbaum FR. Haematopoietic cell transplantation as immunotherapy. Nature. 2001 May 17;411(6835):385-9. doi: 10.1038/35077251. PMID 11357147
- [Background] Amrolia PJ, Muccioli-Casadei G, Yvon E, Huls H, Sili U, Wieder ED, Bollard C, Michalek J, Ghetie V, Heslop HE, Molldrem JJ, Rooney CM, Schlinder J, Vitetta E, Brenner MK. Selective depletion of donor alloreactive T cells without loss of antiviral or antileukemic responses. Blood. 2003 Sep 15;102(6):2292-9. doi: 10.1182/blood-2002-11-3516. Epub 2003 May 22. PMID 12763937
- [Background] Andre-Schmutz I, Le Deist F, Hacein-Bey-Abina S, Vitetta E, Schindler J, Chedeville G, Vilmer E, Fischer A, Cavazzana-Calvo M. Immune reconstitution without graft-versus-host disease after haemopoietic stem-cell transplantation: a phase 1/2 study. Lancet. 2002 Jul 13;360(9327):130-7. doi: 10.1016/S0140-6736(02)09413-8. PMID 12126823
- [Result] Mielke S, McIver ZA, Shenoy A, Fellowes V, Khuu H, Stroncek DF, Leitman SF, Childs R, Battiwalla M, Koklanaris E, Haggerty J, Savani BN, Rezvani K, Barrett AJ. Selectively T cell-depleted allografts from HLA-matched sibling donors followed by low-dose posttransplantation immunosuppression to improve transplantation outcome in patients with hematologic malignancies. Biol Blood Marrow Transplant. 2011 Dec;17(12):1855-61. doi: 10.1016/j.bbmt.2011.05.019. Epub 2011 May 31. PMID 21684344
- [Derived] McIver ZA, Yin F, Hughes T, Battiwalla M, Ito S, Koklanaris E, Haggerty J, Hensel NF, Barrett AJ. Second hematopoietic SCT for leukemia relapsing after myeloablative T cell-depleted transplants does not prolong survival. Bone Marrow Transplant. 2013 Sep;48(9):1192-7. doi: 10.1038/bmt.2013.39. Epub 2013 Mar 25. PMID 23524640
- [Derived] Melenhorst JJ, Tian X, Xu D, Sandler NG, Scheinberg P, Biancotto A, Scheinberg P, McCoy JP Jr, Hensel NF, McIver Z, Douek DC, Barrett AJ. Cytopenia and leukocyte recovery shape cytokine fluctuations after myeloablative allogeneic hematopoietic stem cell transplantation. Haematologica. 2012 Jun;97(6):867-73. doi: 10.3324/haematol.2011.053363. Epub 2011 Dec 1. PMID 22133778
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-H-0136.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Selective T Cell Depletion Transplant Recipients: Subjects will receive a myeloablative conditioning regimen of cyclophosphamide, fludarabine and total body irradiation, followed by an infusion of a stem cell product prepared using the Miltenyi CliniMacs system for CD34 selection and a lymphocyte product that has been selectively depleted using the photodepletion approach. Older subjects will receive a lower dose of irradiation to reduce the regimen intensity. To determine appropriate level of post transplant immunosuppression, a three sequential de-escalation stage design for timing of cyclosporine will be utilized.
Period: Overall Study
Arm/Group | Selective T Cell Depletion Transplant Recipients
Started | 31
Completed | 24
Not Completed | 7
Not completed — Technical Failures | 5
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Selective T Cell Depletion Transplant Recipients
Number analyzed (Participants) | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 3

OUTCOME MEASURES:

1. Primary Outcome: To Determine if Selective T Cell Depletion Using the Photodepletion Procedure Can Substantially Reduce the Rate of Severe Acute GVHD (Grade III/IV) After Matched Sibling Transplantation Followed by Low-dose or no Immunosuppression.
Description: Patients will receive a selectively photodepleted lymphocyte product which will be delivered together with the T cell depleted stem cell product on the day of transplantation. Subjects will receive a conditioning regimen of cyclophosphamide, fludarabine and total body irradiation followed by an infusion of a stem cell product prepared using the Miltenyi CliniMacs system for CD34-selection and a lymphocyte product that has been selectively depleted using the photodepletion approach. Older subjects will receive a lower dose of irradiation to reduce the regimen intensity. To determine appropriate level of post transplant immunosuppression, a three sequential de-escalation stage design for timing of cyclosporine will be utilized. To determine if selective T cell depletion using the photodepletion procedure can substantially reduce the number of severe acute GVHD (grade III/IV) after transplantation followed by low-dose or no immunosuppression.
Time Frame: Day 90
Population: The study accrued 31 transplant recipents and 30 donors. Of the 31 transplant recipients, there were 24 evaluable recipients. Seven of the 24 recipients did not receive transplantation.
Measure: Number; unit: participants
Groups:
- Selective T Cell Depletion Transplant Recipients: Subjects will receive a myeloablative conditioning regimen of cyclophosphamide, fludarabine and total body irradiation, followed by an infusion of a stem cell product prepared using the Miltenyi CliniMacs system for CD34 selection and a lymphocyte product that has been selectively depleted using the photodepletion approach (Kiadis Pharma). Older subjects will receive a lower dose of irradiation to reduce the regimen intensity.
  To determine appropriate level of post transplant immunosuppression.
Arm/Group | Selective T Cell Depletion Transplant Recipients
Number analyzed (Participants) | 24
participants
  Subjects affected by Acute Grade III/ IV GVHD | 3
  Subjects unaffected by Acute Grade III/ IV GVHD | 21

ADVERSE EVENTS:
Arm/Group | Selective T Cell Depletion Transplant Recipients
Serious Adverse Events (participants affected / at risk) | 24/31
Other Adverse Events (participants affected / at risk) | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selective T Cell Depletion Transplant Recipients (N=31)
Infection with normal absolute nuetrophil count (Infections and infestations) | 3 (3)
Infection (Infections and infestations) | 12 (12)
Infection with cytomegalovirus reactivation (Infections and infestations) | 3 (3)
Febrile neutropenia (Infections and infestations) | 1 (1)
Infection with neutropenic fever (Infections and infestations) | 7 (7)
Infection cytomegalovirus gastritis (Infections and infestations) | 1 (1)
pulmonary infection (Infections and infestations) | 1 (1)
renal infection (Infections and infestations) | 1 (1)
multiple opportunistic infection (Infections and infestations) | 1 (1)
GVHD (Immune system disorders) | 6 (6)
GVHD/ infection (Immune system disorders) | 1 (1)
GVHD/ gastrointestinal (Immune system disorders) | 3 (3)
GVHD/ neurology (Nervous system disorders) | 1 (1) — Seizures
GVHD/ pulmonary (Immune system disorders) | 1 (1) — interstitial pneumonitis
GVHD/ cytomegalovirus reactivation (Immune system disorders) | 1 (1)
Disease progression/ Infection (Blood and lymphatic system disorders) | 1 (1)
Adbdominal mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Disease relapse (Blood and lymphatic system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No